CLINICAL TRIAL: NCT01281644
Title: Treatment of Keratosis Pilaris With 810 nm Diode Laser
Acronym: KP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Associate Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA111810
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Keratosis Pilaris (KP)
Keywords: Keratosis pilaris (KP)
MeSH Terms: conditions — Burnett Schwartz Berberian syndrome | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Laser Treatment (No Intervention)
- 45-60 J Diode Laser Therapy (Active Comparator): Diode laser therapy will be initiated at 45-60 J for 30 ms to 100 ms.
  Interventions: Device: Diode Laser

INTERVENTIONS:
Device: Diode Laser — 810 nm diode laser
  Arms: 45-60 J Diode Laser Therapy

SUMMARY:
The investigators hope to establish whether or not the diode laser, a longer-wavelength laser, is effective in treating keratosis pilaris, and hopefully opening a door into the discussion and management of this skin condition. The primary outcome of interest is the difference in the overall blind rater severity scores of the treated versus the untreated sites. The secondary outcome of interest is the change in the patient's self-rated severity score of the treated site. To account for potential natural disease progression or regression, the investigators will also compare patient mean changes to the mean changes in severity scores of the untreated site.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age 18 to 65
* Subject has diagnosis of keratosis pilaris involving both arms
* Subject has Fitzpatrick Skin Type I - III
* Subject is in good health
* Subject has the willingness and ability to understand and provide informed consen

Exclusion Criteria:

* Under 18 or over 65 years of age
* Subjects with Fitzpatrick Skin Type greater than III
* Subjects who have received any laser therapy to the armsin the past year
* Subjects with concurrent diagnosis of another skin condition or malignancy
* Subjects with tan or sunburn over the upper arms in the past month
* Subjects with open, non-healing sores or infections at any skin site
* Subjects who are unable to understand the protocol or give informed consent
* Subjects who take oral photosensitizing medications or who apply topical photosensitizing medications to either arm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Ibrahim O, Khan M, Bolotin D, Dubina M, Nodzenski M, Disphanurat W, Kakar R, Yoo S, Whiting D, West DP, Poon E, Veledar E, Alam M. Treatment of keratosis pilaris with 810-nm diode laser: a randomized clinical trial. JAMA Dermatol. 2015 Feb;151(2):187-91. doi: 10.1001/jamadermatol.2014.2211. PMID 25372313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The principal investigator selected patients presenting to the Dermatology Clinic at Northwestern Memorial Hospital who met the inclusion criteria. A brief, written description of the study was given to the patient.
Groups:
- Subjects Receiving Split Body Treatment: The unit of randomization was the individual arm within each subject to receive either laser therapy on the right arm or on the left arm.
  Each subject received treatment using the 810 nm pulsed diode laser to the arm randomized to be the treatment site.
Period: Overall Study
Arm/Group | Subjects Receiving Split Body Treatment
Started | 23
Completed | 18
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Receiving Split Body Treatment
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Difference in Disease Severity Scores
Description: The primary outcome measure was the difference in disease severity total score, combining redness and roughness/bumpiness scales, between the treated site and the control site, as rated by the blinded dermatologists at 12 weeks post-initial visit. These scales were not validated, as no relevant validated scale was available. However, raters were trained and calibrated on the use of the scale, and prior to review of study images, were asked to rate archival skin images on the same 4-point qualitative subscales used in the study. Each scale ranged from 0 to 3, with 0 being none and 3 being severe. The total score summed the redness and roughness/bumpiness scale scores for a range of 0 (none/better outcome) to 6 (severe/worse outcome).
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Units Other Than Participants: Arm
Arm/Group | No Laser Treatment | 45-60 J Diode Laser Therapy
Number analyzed (Participants) | 18 | 18
Number analyzed (Arm) | 18 | 18
units on a scale | 4 [3 to 5] | 3 [2 to 4]

2. Secondary Outcome: Patient Self-rated Severity
Description: This outcome measure was the difference in disease severity total score, combining redness and roughness/bumpiness scales, between the treated site and the control site, as rated by the patient at 12 weeks post-initial visit. These scales were not validated, as no relevant validated scale was available. Each scale ranged from 0 to 3, with 0 being none and 3 being severe. The total score summed the redness and roughness/bumpiness scale scores for a range of 0 (none/better outcome) to 6 (severe/worse outcome).
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Units Other Than Participants: arms
Arm/Group | No Laser Treatment | 45-60 J Diode Laser Therapy
Number analyzed (Participants) | 18 | 18
Number analyzed (arms) | 18 | 18
units on a scale | 4 [3 to 4] | 2.5 [2 to 4]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | No Laser Treatment | 45-60 J Diode Laser Therapy
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Laser Treatment (N=23) | 45-60 J Diode Laser Therapy (N=23)
post-inflammatory hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes